CLINICAL TRIAL: NCT05434559
Title: Evaluation of Glycemic Control in Adults With Type 1 Diabetes When Switching to Insulin Degludec: a Retrospective Study
Brief Title: Evaluation of Glycemic Control in Adults With Type 1 Diabetes When Switching to Insulin Degludec
Acronym: GLADE
Status: Completed | Type: Observational
Sponsor: prof dr Pieter Gillard (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor-Investigator, prof dr Pieter Gillard, Coordinating Investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: S66239
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Degludec; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: People with type 1 diabetes who switched to Insulin Degludec from another basal insulin between 1/5/2019 and 1/6/2021 in the two participating sensors
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: Insulin Degludec — Switch during standard routine care to Insulin Degludec.

SUMMARY:
Retrospective multicenter study analyzing data gathered from medical records and diabetes management platforms to assess the effect of using Insulin Degludec (Tresiba®) on measures of diabetes control.

People with type 1 diabetes who switched to Insulin Degludec from another basal insulin between 1/5/2019 and 1/6/2021 will be included.

Glycemic control from 12 months before the switch to Insulin Degludec will be compared to glycemic control of the 12 months after the switch.

ELIGIBILITY:
Inclusion Criteria:

* People with T1D ≥18 years at the moment of switch to Insulin Degludec
* Diagnosed with T1D ≥2 years before switch to Insulin Degludec
* On basal-bolus insulin therapy with insulin pens ≥2 years before switch to Insulin Degludec
* ≥6 months use of Insulin Degludec at moment of datacollection
* Using continuous glucose monitoring ≥2 years before switch to Insulin Degludec

Exclusion Criteria:

* People with T1D <18 years at the moment of switch to Insulin Degludec
* People without T1D or with T1D <2 years before switch to Insulin Degludec
* Women with T1D who are pregnant or planning pregnancy during -12 and +12 months
* Not using basal-bolus insulin therapy with insulin pens during -24 and +6 months
* Start to use non-insulin antidiabetic agents between -12 and +12 months
* Having received treatment with oral or injectable corticosteroids during -12 and +12 months
* Undergoing hemodialysis, renal transplantation, or beta cell transplantation during -12 and +12 months
* <6 months use of Insulin Degludec at moment of datacollection
* Not using continuous glucose monitoring or <2 years before switch to Insulin Degludec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every person who meet the inclusion criteria and who is/was followed at the two participating centers during the sampling period will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Time in range | 12 months
  the change in time in range (TIR: 70-180 mg/dL, averaged per month) over 24 hours between 12 (±2) months before switch to 12 (±2) months after switch to Insulin Degludec

SECONDARY OUTCOMES:
HbA1c | 12 months
  difference in HbA1c between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Time below 54 mg/dL | 12 months
  difference in time in clinically significant hypoglycemia (<54 mg/dL averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Time in range | 12 months
  difference in TIR (70-180 mg/dL, averaged per month) from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Time below 70 mg/dL | 12 months
  difference in time below range (<70 mg/dL averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Time above 180 mg/dL | 12 months
  difference in time above range (>180 mg/dL averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Time above 250 mg/dL | 12 months
  difference in time in significant hyperglycemia (>250 mg/dL averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Mean glucose | 12 months
  difference in mean glucose (averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Glycemic variability | 12 months
  difference in glycemic variability (standard deviation, coefficient of variation; averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Insulin dose | 12 months
  difference in insulin dose (total daily dose, basal dose, bolus dose) between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Body mass index | 12 months
  difference in body mass index (BMI) between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec

OTHER OUTCOMES:
Hospital visits and/or admissions due to hypoglycemia or ketoacidosis | 12 months
  difference in number of hospital visits and/or admissions due to hypoglycemia or ketoacidosis between 12 [±2] months before switch to 12 [±2] months after switch to Insulin Degludec
Participants who discontinue the use of Insulin Degludec | 12 months
  number of participants who discontinue the use of Insulin Degludec
Reason for discontinuation of Insulin Degludec | 12 months
  overview of reasons to discontinue Insulin Degludec (in tabular view)
Indication for use of Insulin Degludec | baseline
  overview of reasons to start Insulin Degludec (in tabular view)
Glycemic consensus targets | 12 months
  proportion of people reaching HbA1c and glucose consensustargets 12 [±2] months after switch to Insulin Degludec

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven
  - University Hospital Antwerp, Wilrijk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Groote R, Lefever E, Charleer S, Donne P, De Block C, Mathieu C, Gillard P. Continuous Glucose Monitoring-Derived Glucometrics in Adults with Type 1 Diabetes When Switching Basal Insulins. Diabetes Technol Ther. 2024 Aug;26(8):587-595. doi: 10.1089/dia.2023.0616. Epub 2024 Apr 9. PMID 38512387